CLINICAL TRIAL: NCT00053365
Title: A Phase II Evaluation Of Irofulven (IND #55804, NSC #683863) In The Treatment Of Recurrent Or Persistent Platinium-Sensitive Ovarian Or Primary Peritoneal Cancer
Brief Title: Irofulven in Treating Patients With Recurrent or Persistent Ovarian Epithelial or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02512; NCI-2012-02512 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000269484; GOG-0146O (Other: Gynecologic Oncology Group); GOG-0146O (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — irofulven

ARMS (1):
- Treatment (irofulven) (Experimental): Patients receive irofulven IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.
  Interventions: Drug: irofulven

INTERVENTIONS:
Drug: irofulven — Given IV
  Other Names: 6-hydroxymethylacylfulvene; HMAF; MGI 114; MGI-114

SUMMARY:
Phase II trial to study the effectiveness of irofulven in treating patients who have recurrent or persistent ovarian epithelial cancer or primary peritoneal cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the antitumor activity of irofulven in patients with persistent or recurrent platinum-sensitive ovarian epithelial or primary peritoneal cancer.

II. Determine the toxicity of this drug in these patients.

OUTLINE:

Patients receive irofulven IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression.

Patients are followed at approximately 30 days, every 3 months for 2 years, and then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 22-60 patients will be accrued for this study within at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal carcinoma

  * Recurrent or persistent disease
* At least 1 unidimensionally measurable target lesion* defined as:

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Must have received 1 prior platinum-based chemotherapeutic regimen containing carboplatin, cisplatin, or another organoplatinum compound for primary disease

  * Initial treatment may have included high-dose, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * Patients who have not received prior paclitaxel may receive a second regimen containing paclitaxel
* Ineligible for a higher priority GOG protocol (e.g., any active phase III GOG protocol for the same patient population)
* Platinum-sensitive disease

  * Platinum-free interval** of more than 6 months, but less than 12 months duration, with no clinical evidence of progressive disease after response to platinum
* Performance status - GOG 0-2 for patients who received 1 prior therapy regimen
* Performance status - GOG 0-1 for patients who received 2 prior therapy regimens
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No prior congestive heart failure requiring medication
* No uncontrolled hypertension within the past 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer
* No history of retinopathy and/or macular degeneration
* No neuropathy (sensory and motor) greater than grade 1
* No active infection requiring antibiotics
* No other illness or condition that would preclude study entry
* No prior bone marrow or stem cell transplantation
* At least 3 weeks since prior biologic therapy or immunotherapy for malignant tumor
* One prior non-cytotoxic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule signal transduction inhibitors) allowed
* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No prior irofulven
* No additional prior cytotoxic chemotherapy for recurrent or persistent disease, including retreatment with initial chemotherapy regimens
* At least 1 week since prior hormonal therapy for malignant tumor
* Concurrent hormone replacement therapy allowed
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas
* Recovered from recent prior surgery
* At least 3 weeks since any other prior therapy for malignant tumor
* No prior anticancer treatment that would preclude study therapy
* One prior noncytotoxic cytostatic regimen for recurrent or persistent disease allowed

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schilder, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stage I of the study accrued patients from 6/2/2003 through 10/31/2005. Stage II of the study accrued patients from 1/3/2006 through 4/7/2008.
Period: Overall Study
Arm/Group | Treatment (Irofulven)
Started | 61
Completed | 55
Not Completed | 6
Not completed — Incorrect cell type | 1
Not completed — Platinum-sensitive interval >12 months | 1
Not completed — Never treated | 4

BASELINE CHARACTERISTICS:
Population: This is the number of eligible and evaluable participants.
Arm/Group | Treatment (Irofulven)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.7)
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 10
  50-59 years | 17
  60-69 years | 21
  70-79 years | 4
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Recurrent/Persistent Disease [Number; unit: participants] — FIGO (International Federation of Gynecology and Obestetrics) Stage Grouping for Primary Carcinoma of the Ovary(1985)
  participants | 55
Cell Type [Number; unit: participants]
  Endometrioid Adenocarcinoma | 2
  Mixed Epithelial Carcinoma | 3
  Serous Adenocarcinoma | 47
  Undifferentiated Carcinoma | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Per Gynecologic Oncology Group(GOG) Response Evaluation Criteria in Solid Tumors(RECIST) Criteria: Complete Response is disappearance of all target and non-target lesions; Partial Response is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable dimensions; Increasing Disease is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Response is to be evaluated every 42 days for the first 6 months and every 6 months thereafter while the patient is receiving study treatment, then every 3 months for 2 years and every 6 months for the next 3 years until documented progression or death.
Time Frame: From entry into study until documented progression or death, assessed up to 5 years.
Measure: Number; unit: participants
Arm/Group | Treatment (Irofulven)
Number analyzed (Participants) | 55
participants
  Partial Response | 7 [0.07 to 0.29]
  Stable Disease | 30
  Increase Disease | 12
  Indeterminate | 6

2. Primary Outcome: Frequency and Severity of Observed Adverse Events, Grade 3 or Higher According to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and evaluable patients
Measure: Number; unit: participants
Groups:
- Grade 3 (CTCAE v 2.0): Number of patients who experienced a grade 3 event using Common Toxicity Criteria version 2.0
- Grade 4 (CTCAE v 2.0): Number of patients who experienced a grade 4 event using Common Toxicity Criteria version 2.0
Arm/Group | Grade 3 (CTCAE v 2.0) | Grade 4 (CTCAE v 2.0)
Number analyzed (Participants) | 55 | 55
participants
  Leukopenia | 11 | 0
  Thrombocytopenia | 11 | 2
  Neutropenia | 16 | 6
  Other hematologic | 6 | 0
  Constitutional | 4 | 0
  Gastrointestinal | 8 | 1
  Infection | 4 | 0
  Musculoskeletal | 2 | 0
  Metabolic | 2 | 1
  Neuropathy (sensory) | 1 | 0
  Other neurologic | 2 | 0
  Ocular | 4 | 0
  Pain | 1 | 0

3. Secondary Outcome: Progression-free Survival
Description: Per Gynecologic Oncology Group(GOG) Response Evaluation Criteria in Solid Tumors(RECIST) Criteria, progression is defined as at least a 20% increase in the sum of longest dimesions(LD) of target lesions taking as reference the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
Time Frame: From entry into study to death or date of last contact, assessed up to 5 years
Population: Eligible and evaluable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Irofulven)
Number analyzed (Participants) | 55
months
  Median Overall Survival | 24.1 [17.5 to 28.9]
  Median Progression-free Survival | 6.7 [4.1 to 8.9]

ADVERSE EVENTS:
Time Frame: Adverse Events(AEs) considered to be due to study treatment are to be reported up until 5 years after initiating treatment.
Description: A patient's AEs are reported following each cycle of study treatment and include AEs occurring within 30 days of each cycle.
Arm/Group | Treatment (Irofulven)
Serious Adverse Events (participants affected / at risk) | 18/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Irofulven) (N=55)
Cardiovascular Other (Cardiac disorders) | 1
Thrombosis Embolism (Cardiac disorders) | 1
Anorexia (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 2
Vomitting (Gastrointestinal disorders) | 3
Gi Other (Gastrointestinal disorders) | 2
Infection Without Neutropenia (Infections and infestations) | 2
Hypomagnesmia (Metabolism and nutrition disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Ataxia(Incoordination) (Nervous system disorders) | 3
Neuropathy Sensor (Nervous system disorders) | 1
Ocular Other (Eye disorders) | 1
Vision Photophobia (Eye disorders) | 2
Vision Blurres (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Irofulven) (N=55)
Neutropenia (Blood and lymphatic system disorders) | 38
Thrombocytopenia (Blood and lymphatic system disorders) | 41
Lymphopenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 39
Transfusion Prbc's (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 45
Sinus Tachycardia (Cardiac disorders) | 3
Edema (Cardiac disorders) | 5
Fever(No Neutropenia) (General disorders) | 4
Sweating (General disorders) | 3
Fatigue (General disorders) | 41
Pruritis (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10
Rash Desquamation (Skin and subcutaneous tissue disorders) | 5
Bruising (Skin and subcutaneous tissue disorders) | 3
Hot Flashes/Flushes (Endocrine disorders) | 7
Anorexia (Gastrointestinal disorders) | 12
Flatulence (Gastrointestinal disorders) | 6
Dyspepsia/Heartburn (Gastrointestinal disorders) | 10
Dysphagia Esophagitis Odynophagia (Gastrointestinal disorders) | 4
Diarrhea Without Colostomy (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 22
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 7
Vomitting (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 38
Hematuria No Vaginal Bleeding (Vascular disorders) | 3
Hypoalbuminemia (Hepatobiliary disorders) | 5
Sgot(Alt) (Hepatobiliary disorders) | 7
Sgot(Ast) (Hepatobiliary disorders) | 5
Alkaline Phosphatase (Hepatobiliary disorders) | 6
Infection Without Neutropenia (Infections and infestations) | 9
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesmia (Metabolism and nutrition disorders) | 10
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 3
Ataxia(Incoordination) (Nervous system disorders) | 3
Insomnia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 7
Mood Alteration Depression (Nervous system disorders) | 4
Neuropathy Sensor (Nervous system disorders) | 19
Ocular Other (Eye disorders) | 5
Dry Eye (Eye disorders) | 3
Vision Photophobia (Eye disorders) | 5
Vision Flashing Lights/Floaters (Eye disorders) | 9
Vision Blurres (Eye disorders) | 8
Abdominal Pain (General disorders) | 18
Pain Other (General disorders) | 7
Headache (General disorders) | 17
Arthralgia (General disorders) | 3
Myalgia (General disorders) | 8
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Urinary Retention (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less